CLINICAL TRIAL: NCT06056284
Title: The Effect of Progressive Relaxation Exercise and Sleep Hygiene Training on Sleep Quality and AnxietyLevel Given to Outpatients With Anxiety Disorder in Psychiatry Outpatient Clinic
Brief Title: The Effect of Progressive Relaxation Exercise and Sleep Hygiene Training on Sleep Quality and AnxietyLevel Given to Outpatients With Anxiety Disorder in Psychiatry Clinic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Nur Eda Bal, investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SaglikBilimleriU-SBE-NEB-01
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Anxiety Disorder/Anxiety State
Keywords: Sleep hygiene; Anxiety; progressive relaxation exercise; anxiety disorder
MeSH Terms: conditions — Anxiety Disorders; Sleep Hygiene

STUDY DESIGN:
Intervention Model Description: two groups with experimental and control group
Who Masked: Participant, Outcomes Assessor
Masking Description: The experimental group will be subjected to progressive relaxation exercise and the outcome assesment will be performend by an outcomes assessor blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive relaxation exercise and sleep hygiene training (Experimental): It is planned to include 26 patients in the experimental group. Voluntary Consent Form, Personal Information Form, Pittsburgh Sleep Quality Index (PSQI), Sleep Hygiene Index (SHI) and Beck Anxiety Scale (BAS) will be applied to the patients in the experimental group in the first week of the 7-week study. Data will be collected by face-to-face interviews with the patients and an appointment will be made for the post-test after seven weeks. In the second week, the individuals in the experimental group will be taught progressive relaxation exercise in the hospital environment by the researcher using the compact disc (CD) prepared by the Turkish Psychological Association and after the sleep hygiene training, the progressive relaxation exercise brochure and sleep hygiene training brochure created by the researcher will be distributed. As of the second week, the individuals in the experimental group will be expected to apply the trainings given twice in the hospital environment.
  Interventions: Behavioral: Progressive relaxation exercises and sleep hygiene training
- Control group (No Intervention): It is planned to include 26 patients in the control group. Voluntary Consent Form, Personal Information Form, Pittsburgh Sleep Quality Index (PSQI), Sleep Hygiene Index (SHI) and Beck Anxiety Scale (BAS) will be applied to the individuals in the control group in the first week of the 7-week research programme. Data will be collected by face-to-face interview with the patients. Individuals in the control group will not be given any training by the researcher. Individuals in the control group will be given an appointment for the post-test after seven weeks. At the end of seven weeks, individuals in the control group will be asked to fill in the Pittsburgh Sleep Quality Index (PSQI), Sleep Hygiene Index (SHI) and Beck Anxiety Scale (BAS) again.

INTERVENTIONS:
Behavioral: Progressive relaxation exercises and sleep hygiene training — Voluntary Consent Form, Personal Information Form, Pittsburgh Sleep Quality Index (PSQI), Sleep Hygiene Index (SHI) and Beck Anxiety Scale (BAS) will be applied to the patients in the experimental group in the first week of the 7-week study. Data will be collected by face-to-face interviews with the patients. After seven weeks, an appointment will be given for the post-test. In the second week, those in the experimental group will be taught progressive relaxation exercise using a compact disc (CD) prepared by the Turkish Psychological Association in the hospital and after the sleep hygiene training, progressive relaxation exercise brochure and sleep hygiene training brochure will be distributed. Starting from the second week, the individuals in the experimental group will be expected to apply the trainings given in the hospital accompanied by the researcher two days a week for six weeks and to apply the trainings given to the individuals at home on the other days of the week.
  Arms: Progressive relaxation exercise and sleep hygiene training

SUMMARY:
The aim of this study was to investigate the effect of progressive relaxation exercise and sleep hygiene training on sleep quality and anxiety levels in patients diagnosed with anxiety disorder admitted to psychiatry outpatient clinic.

DETAILED DESCRIPTION:
The population of the study consisted of 1417 patients diagnosed with anxiety disorder who applied to the psychiatry outpatient clinic of Ankara Kızılcahamam State Hospital between December 2021 and February 2022. For the pretest-posttest control group research, the required sample size was determined as 47 using the G*Power 3.1.9.4 program with 95% power based on Cohen's d = 0.5 medium effect size alpha = 0.05. However, considering the data loss that may occur in the study, the sample size was determined as 52 when the dropout rate was determined as 10%. The age range of the research sample is 18-75 years old. Individuals who agree to participate in the study and meet the inclusion criteria will be assigned to the experimental and control groups by simple random sampling method. It is planned to include 26 patients in both the experimental and control groups. In the first week of this 8-week research program, the individuals in the experimental and control groups will be administered the Voluntary Consent Form, Personal Information Form consisting of 17 questions prepared by the researcher by reviewing the literature, Pittsburgh Sleep Quality Index (PSQI), Sleep Hygiene Index (SHI) and Beck Anxiety Scale (BAS). Data will be collected by face-to-face interviews with the patients. Individuals in the experimental and control groups will be given an appointment for the posttest eight weeks later. In the second week, individuals in the experimental group will be given sleep hygiene training and a sleep hygiene brochure prepared in line with the literature. In addition, a compact disc (CD) prepared by the Turkish Psychological Association and a training brochure developed by the researcher in line with the progressive relaxation exercises CD, which includes the steps of progressive relaxation exercise application, will be used to teach the progressive relaxation exercise.

The first part of the CD includes a 10-minute description of deep relaxation, its purpose and information to be considered during the exercise. In the second 30-minute part, relaxation exercises are explained with the sound of a stream and verbal instructions. The last 30-minute section included only relaxation music without audio instructions. Before the application, each patient in the experimental group will be taught the correct breathing technique by explaining the importance of heavy, deep and quiet breathing. As of the third week, progressive relaxation exercises will be applied to six different patients in groups of two in the hospital environment once a week in three sessions during the day for a total of six weeks with the researcher. In addition, the patients will be expected to repeat the progressive relaxation exercises in their home environment two days a week and will be asked to fill out follow-up charts. The individuals in the control group will not be given any training by the researcher. At the end of eight weeks, the individuals in the experimental and control groups will be asked to fill in the Pittsburgh Sleep Quality Index (PSQI), Sleep Hygiene Index (SHI) and Beck Anxiety Scale (BAS) again. Trainings and administration of the forms will be conducted in an empty room allocated for the researcher.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18 and 60
* Having been diagnosed with anxiety disorder at least 6 months ago
* No barriers in Turkish oral and written communication
* Volunteering to participate in the research
* Not having received progressive relaxation exercise and sleep hygiene training before
* To reside in Kızılcahamam district centre
* Not having Chronic Obstructive Pulmonary Disease (COPD), Heart Failure, asthma, Musculoskeletal System Diseases, etc. which may prevent progressive relaxation exercise

Exclusion Criteria:

* The individual has conditions that impair the ability to assess reality, such as psychosis, being in the manic phase of bipolar disorder
* Chronic Obstructive Pulmonary Disease (COPD), Heart Failure, asthma, Musculoskeletal System Diseases, etc. that may prevent progressive relaxation exercise
* The individual has participated in another progressive relaxation exercise and/or sleep hygiene training programme
* The individual is taking a psychiatric drug with a relaxant effect

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Beck Anxiety Scale (BAS) | seven weeks
  Developed in 1988, its Turkish validity and reliability was performed by Ulusoy et al. (1998) and cronbach alpha was found to be 0.93. It is a 4-point Likert-type scale consisting of 21 questions aiming to measure the severity of anxiety of the individual. Each question is scored between 0-3. The total score obtained from the scale indicates low level of anxiety if the score is between 8-15 points, moderate level of anxiety if the score is between 16-25 points, and high level of anxiety if the score is between 26-63 points.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | seven weeks
  A PDQI score greater than 5 indicates poor sleep quality. The scale The validity and reliability study in Turkey was conducted by Ağargün et al. in 1996. The Cronbach's alpha reliability coefficient of the scale was 0.804. was found. The sleep quality scale consists of 18 self-report questions and assesses sleep quality in the last 4 weeks. PDQI consists of 18 items and 7 component scores. grouped. Some of the components are indicated by a single item, others are is obtained by combining several items. Each item is scored on a 0-3 point scale. is evaluated. The sum of the 7 component scores has a value between 0-21. Total A high score indicates poor sleep quality.
Sleep Hygiene Index (SHI) | seven weeks
  It was developed by Mastin et al. (2006). Its Turkish validity and reliability was conducted by Özdemir et al. The scale consists of 13 questions and has a five-point Likert scale format (none: 1, rarely: 2, sometimes: 3, often: 4, always: 5). The index is based on the participant's sleep hygiene It aims to assess the presence of sleep hygiene by questioning how often the participant performs sleep behaviors. Scores range from 13 to 65, with higher scores indicating worse sleep hygiene status of the participant. The items that make up the Sleep Hygiene Index are derived from the diagnostic criteria for poor sleep hygiene in the International Classification of Sleep Disorders. The Cronbach Alpha value of the Sleep Hygiene Index was calculated as 0.70 and found to be valid and reliable.

CONTACTS AND LOCATIONS:
Locations (1):
- Kızılcahamam State Hospital, Ankara, Kızılcahamam, Turkey (Türkiye)